CLINICAL TRIAL: NCT01598051
Title: Treatment Satisfaction Under Rivaroxaban (ACTS/TSQM)
Brief Title: Xarelto [SPAF-QOL] Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16296
Record Dates: First submitted 2012-04-20; First posted 2012-05-15 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Xarelto; SPAF; QOL
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients treated with Xarelto under practical manner for SPAF.
  Interventions: Drug: Rivaroxaban (Xarelto_ BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto_ BAY59-7939) — Patients treated with Xarelto under practical manner for SPAF.

SUMMARY:
The objective of this study is to understand if Rivaroxaban can improve treatment satisfaction of Warfarin patients and assess the safety and effectiveness of Xarelto in real clinical practice.

A total of 725 patients are to be enrolled and followed for a 6 months.period. QOL survey will be conducted at month 0, 3, 6 using ACTS/TSQM.

This study is categorized as a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Xarelto for SPAF.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by Warfarin for their atrial fibrillation for at least two months at the time of the study initiation.
* Rivaroxaban naïve patients
* Patients 20 years old or older.
* Patients who agree to sign the inform consent

Exclusion Criteria:

* Patients who are contraindicated by product label

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation necessary for the treatment for prevention of ischemic stroke and systemic embolism
Sampling Method: Non-Probability Sample
Enrollment: 741 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Improvement of treatment satisfaction (Evaluated through ACTS and TSQM questionnaires) | Up to 6 months
Incidence of ADRs and serious AEs (especially for hemorrhagic events, and liver disfunction with increase of liver-function-relating enzymes including bilirubin) | Up to 6 months
Incidence of events of stroke | Up to 6 months
Incidence of events of non-central nervous system embolism | Up to 6 months

OTHER OUTCOMES:
Treatment satisfaction scores at Month 3 and Month 6 by demographic and clinical characteristics | At Month 3 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Background] Koretsune Y, Kumagai K, Uchiyama S, Yamashita T, Yasaka M, Watanabe-Fujinuma E, Banderas BF, Akiyama S, Okayama Y, Briere JB, Dickie G, Cano SJ. Patient-reported treatment satisfaction with rivaroxaban in Japanese non-valvular atrial fibrillation patients: an observational study. Curr Med Res Opin. 2018 Dec;34(12):2157-2164. doi: 10.1080/03007995.2018.1507315. Epub 2018 Aug 14. PMID 30067119
- [Derived] Watanabe-Fujinuma E, Banderas BF, Koretsune Y, Kumagai K, Uchiyama S, Yamashita T, Yasaka M, Akiyama S, Briere JB, Dickie G, Cano SJ. Psychometric validation of anti-clot treatment scale and treatment satisfaction questionnaire for medication version II in Japanese patients with atrial fibrillation. J Med Econ. 2019 Aug;22(8):798-805. doi: 10.1080/13696998.2019.1609003. Epub 2019 May 13. PMID 30995146
- [Derived] Gavrilov SG, Lebedev IS. Is the endovascular embolization of tributaries of the internal iliac veins essential in the treatment of isolated pelvic-perineal reflux? Curr Med Res Opin. 2019 Jan;35(1):27-31. doi: 10.1080/03007995.2018.1498781. Epub 2018 Jul 25. PMID 29985674